CLINICAL TRIAL: NCT06927518
Title: Effects of Receptive Language Intervention vs Individual Therapy for Preschool Children With
Brief Title: Effects of Receptive Language Intervention vs Individual Therapy for Preschool Children With Autism Spectrum Disorder.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0655
Record Dates: First submitted 2025-04-07; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individual Therapy (Experimental): 14 participant will receive individual therapy. Each participant will receive 3 session per week for 2 Months.
  Interventions: Other: Receptive language intervention by using the total communication
- Group Therapy (Active Comparator): 16 participants will divided in 2 groups. each group will receive 3 session per week for 2 Months.
  Interventions: Other: Receptive language intervention by using the total communication

INTERVENTIONS:
Other: Receptive language intervention by using the total communication — Receptive language intervention using Total Communication (TC) for children with autism can be highly effective. Total Communication involves using a combination of communication methods to support language comprehension and expression. It recognizes that individuals with autism often benefit from multi-modal communication rather than relying solely on spoken language.

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder characterized by deficits in social communication and social interaction and the presence of restricted, repetitive behaviors. Atypical behaviors, conditioning, and difficulties interacting with others are emblems of Autism spectrum disorder (ASD). Autism spectrum disorder (ASD) frequently affects receptive language skills essential for comprehension and communication. Early intervention is crucial for optimizing language outcomes. This randomized controlled trial (RCT) investigates the comparative efficacy of receptive language intervention (RLI) in group versus individual therapy settings for preschool children with ASD.

This study aims to investigate the efficacy of receptive language intervention (RLI) in group versus individual therapy settings for preschool children with Autism Spectrum Disorder (ASD) aged 3-5 years. The study aims to address the knowledge gap regarding optimal delivery methods for receptive language interventions. Twenty preschool children (ages 3-5) with ASD will be randomly assigned to either group (n=10) or individual (n=10) therapy conditions. Outcome measures will assess by Laura Mize Teach Me To Talk receptive language checklist, noted before therapy and after completing 20 sessions post-therapy (after 7 weeks). Statistical analysis was done using SPSS 20. An Independent t-test was utilized to see any difference between groups. The study's findings will inform evidence-based practice, enhancing receptive language skills in preschool children with ASD. The study could give precious perceptivity to clinicians, preceptors, and policymakers, helping them make informed, substantiation-based opinions about the most effective and doable intervention strategies. The expected outcomes include comparable receptive language outcomes between group and individual therapy, identification of setting-specific benefits and challenges, and child characteristics influencing treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 5 years diagnosed with ASD.
* Children who are able to attend regular therapy sessions as scheduled in the study (either group or individual therapy).
* Both male and female will be included.

Exclusion Criteria:

* Children with co-occurring severe medical conditions.
* Children who have already received intensive speech and language therapy for receptive language skills within the last 6 months.
* Children with behavioral issues so severe (e.g., aggression, extreme hyperactivity) that they might disrupt group therapy sessions or be unable to focus in individual therapy.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-07-29 (Estimated)

PRIMARY OUTCOMES:
Laura Mize Teach Me To Talk receptive language checklist, Me To Talk receptive language checklist, | 2 months
  Laura Mize, a pediatric speech-language pathologist, created the "Teach Me To Talk" resources, including a Receptive Language Skills Checklist. This checklist is designed to help parents, therapists, and educators assess and track a child's receptive language development, particularly for toddlers and young children with language delays or disorders, including autism.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Mariam Zahra, MS SLP, Principal Investigator — Riphah International University
Locations (1):
- Irum Khara, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gajre MP, Shah M, Pradhan SV, Aseri H. Examining the Impact of Group-Based Social Skills Intervention in Autistic Children Aged Eight to 15 Years. Cureus. 2024 Feb 1;16(2):e53376. doi: 10.7759/cureus.53376. eCollection 2024 Feb. PMID 38435203
- [Background] Akbar RF, Kiyani HS, Saqulain G. Effectiveness of group therapy versus individual therapy in acquisition of pre-linguistic skills in children with expressive language disorders. The Rehabilitation Journal. 2023.